CLINICAL TRIAL: NCT06644976
Title: Bleeding of Patients Using NOAC Anticoagulation Therapy in Proximal Femoral Fracture Internal Fixation Surgery
Brief Title: Monitoring Bleeding of Patients Using NOAC Anticoagulation Therapy in Proximal Femoral Fracture Internal Fixation Surgery Without Waiting. We Measure Bleeding in Surgery and the Levels of Noac Drug in Blood. We Will Try to Compare to Regular Pateints Later
Status: Recruiting | Type: Observational
Sponsor: Meir Hospital, Kfar Saba, Israel (Other)
Responsible Party: Principal Investigator, Maron Talmore, Dr. meron pinchas talmor, Meir Hospital, Kfar Saba, Israel
Other Study IDs: mmc000723
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Osteoperosis; Femoral Neck Fractures; Anticoagulant Therapy
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- early surgery
  Interventions: Procedure: femoral neck CRIF
- late surgery
  Interventions: Procedure: femoral neck CRIF

INTERVENTIONS:
Procedure: femoral neck CRIF — femoral neck fracture CRiF while under noac. no special intervention beside taking blood test for drug levels

SUMMARY:
until today we waited at least 24 hours before surgery of femoral neck fractures in patients who take anticouagolation . in our new reasearch we belive that patients who take NOAC can go under surgery earlier with minimal risk

ELIGIBILITY:
Inclusion Criteria:

above 18 y.o femoral neck fracture NOAC capable of making inform consent primary surgery

-

Exclusion Criteria:

* under 18 y.o
* anti platelet therapy (aspirin is not included)
* creatinine clearance under 50
* active anti cancer therapy
* ITP patients
* non capable of making inform consent
* patients which decide not to proceed with the expeirment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with femoral neck fracture thattake noac and arrive at meir hospital and need surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
bleeding | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Hospital, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No